CLINICAL TRIAL: NCT04615793
Title: Effect of Pilates Exercises on Gross Motor Function and Balance in Children With Diplegic Cerebral Palsy
Brief Title: Effect of Pilates Exercises on Gross Motor Function and Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, hanaa mohsen, lecturer in the deparment of pediatrics and peditaric surgery , faculty of phyical therapy, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002914
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: to Determine the Effect of Pilate's Exercises on Gross Motor Function and Balance
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): The control group will receive flexibility exercises and strength training focusing on the trunk and lower limb muscles, postural control exercise in different positions and different surfaces and general endurance training . Control group will receive intervention in the form of five minutes warm up followed by 12 minutes of walking at their comfortable pace and concluded with a five minutes cool down
- EXPERMINTAL GROUP (Experimental): The experimental group will obtain Pilate exercises, consist of strengthening,stretching and coordinated exercises on lower and trunk muscle
  Interventions: Other: PILATES EXERCISES

INTERVENTIONS:
Other: PILATES EXERCISES — The experimental group will receive Pilates exercises focusing on lower limb strength, flexibility and coordination in addition to exercises given to control group. Exercises or movements were done on a mat, on an exercise ball or in standing position while emphasizing on spinal and pelvic alignment, maintaining core contraction and the rhythm of respiration. All exercises were done for 10 repetitions with a rest period of two minutes before commencing the next exercise, and lasted for about 45 minutes. All the groups will receive the above mentioned interventions thrice in a week for a period of 10 week
  Arms: EXPERMINTAL GROUP

SUMMARY:
the study aimed to asses the effect of Pilate exercise on motor function and balance in diplegic children

ELIGIBILITY:
Inclusion Criteria:

* 7 to 9 years,
* mild spasticity of lower limb
* able to understand and follow instructions

Exclusion Criteria:

* fixed contracture
* visual or respiratory disorders,

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
The Pediatric Balance Scale | pre and after 10 week of intervention, the maximum score is 56, so increase the score indicate improvement
  The PBS is a modified version of the Berg balance scale, which is designed to evaluate balance in children with mild to moderate motor impairment. Fifty-six points is the maximum score . This scale evaluates performance of fourteen activities common in everyday life.

SECONDARY OUTCOMES:
Gross motor function | pre and after 10 week of intervension. increase the percentage indicate improvement
  gross motor function consist of 5 dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Badr Univesity in Cairo (BUC), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided